CLINICAL TRIAL: NCT04999722
Title: Establishment and Preliminary Evaluation of Digital Three Level Linkage Whole Process Diabetes Management System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing Renji Hospital, University of Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021CQSDWRMYYEC-004
Record Dates: First submitted 2021-07-19; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Manage; Mobile app
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Mobile app was used for follow-up
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP group (Active Comparator): Participants with diabetes who had access to a mobile APP
  Interventions: Behavioral: Mobile APP management
- Control Group (Placebo Comparator): Diabetes participants who accepted the traditional management model
  Interventions: Behavioral: Traditional mode of management

INTERVENTIONS:
Behavioral: Traditional mode of management — Traditional model management of Diabetes Mellitus patients
  Arms: Control Group
Behavioral: Mobile APP management — Management of diabetic patients with mobile phone APP
  Arms: APP group

SUMMARY:
This study used Nan'an District of Chongqing, China as a pilot project to improve the comprehensive compliance rate of diabetic patients in China, and reduce the physical and economic harm caused by complications.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 2 diabetes.
2. Aged 18-70;
3. HbA1c ≥ 8.0%

Exclusion Criteria:

1. Pregnancy;
2. Chronic kidney disease (CKD stage 5);
3. Senile dementia patients;
4. With malignant tumor;
5. Moderate and severe anemia;
6. Severe liver dysfunction;
7. Hemolytic anemia, aplastic anemia, massive blood loss or transfusion, chronic malaria;
8. In the recent one week, large doses of salicylate, erythropoietin, antiretroviral drugs, ribavirin and other drugs that have an impact on the detection of glycosylated hemoglobin were used

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-08-25 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-24 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Glycated hemoglobin at 12 months | Month 12
  Changes of glycated hemoglobin （percentage）before and after management

SECONDARY OUTCOMES:
Change from Baseline Blood pressure at 12 months | Month 12
  Changes of blood pressure（mmHg） before and after management
Change from Baseline blood lipid at 12 months | Month 12
  Changes of blood lipid （mmol/L）before and after management
Change from Baseline Diabetic nephropathy at 12 months | Month 12
  Changes of Diabetic nephropathy（ratio） before and after management